CLINICAL TRIAL: NCT06595992
Title: EVOLUTION: Prospective Observational Cohort Study of Moderate Aortic Valve Disease
Brief Title: Prospective Observational Cohort Study of Moderate Aortic Valve Disease
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0357
Record Dates: First submitted 2024-08-30; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Moderate Aortic Valve Stenosis; Moderate Aortic Valve Regurgitation; Aortic Valve Disease
Keywords: Aortic Valve Disease Progression; Mortality; Heart Failure
MeSH Terms: conditions — Aortic Valve Disease; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The patient's blood sample is kept in a suitable way, centrifuged and aliquoted, etc., and stored in a -80° freezer。
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this research is to evaluate and predict the progression of moderate aortic stenosis and regurgitation from clinical characterization, biological, echocardiographic, and computed tomography (CT) et. al. Additionally, try to analyze the potential impact of device or drug therapy on the progression of the conditions.

DETAILED DESCRIPTION:
This study is a prospective observational cohort study aimed at thoroughly investigating the disease progression and influencing factors of patients with moderate aortic valve disease, diagnosed at the Second Affiliated Hospital of Zhejiang University School of Medicine. Aortic valve stenosis and aortic regurgitation are the most common forms of aortic valve disease. According to the 2021 ESC guidelines, moderate aortic stenosis (Moderate AS) is defined as an aortic valve area (AVA) of 1.0-1.5 cm2 on echocardiography (or AVA <1.0 cm2 with an AVA index of 0.60-0.85 cm2/m2), a peak jet velocity (Vmax) of 3-4 m/s, and/or a mean transvalvular gradient (MG) of 20-40 mmHg. Moderate aortic regurgitation (Moderate AR) is defined as a regurgitant fraction between 30% and 50% or an effective regurgitant orifice area between 0.10-0.30 cm2.

While treatment guidelines for patients with severe AS are well-established, there is currently no clear consensus on the treatment of patients with moderate AS, and the subsequent disease progression for these patients remains unclear. Similarly, when the aortic valve shows only moderate regurgitation, surgical treatment is usually not required; the most important aspect is regular monitoring of disease changes, including regular echocardiographic examinations. It is noteworthy that the time span from moderate to severe aortic regurgitation can vary from 1 to 10 years, and the monitoring and early warning mechanisms for potential markers indicating disease deterioration are currently not well developed. The goal of this study is to identify all clinical characterization, biological, echocardiographic, and CT imaging parameters that may increase the risk of disease progression. The confirmation of these parameters will guide future research to develop medical and interventional treatment methods to reduce mortality associated with this disease. Patients participating in this study will undergo outpatient follow-up every 1 year after diagnosis and will undergo electrocardiography, echocardiography, blood analysis, and enhanced CT examinations at 1, 3, and 5 years (plus once if an endpoint event occurs). Through these comprehensive monitoring methods, we expect to more accurately assess changes in the patient's condition and provide a scientific basis for clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Be willing and able to provide informed consent to participate in the study
* Patient has moderate aortic valve diseases with echocardiographically derived criteria

Exclusion Criteria:

* Severe aortic valve diseases with echocardiographically derived criteria or planned cardiac surgery or likely need for surgery within 6 months
* Patients who have undergone elective transfemoral transcatheter aortic valve replacement
* Life expectancy is less than 12 months due to non-heart disease (such as cancer, chronic liver disease, chronic kidney disease, or chronic end-stage lung disease, etc.)
* Severe dementia (cannot sign research informed consent, cannot take care of themselves or complete the study visit)
* Acute pulmonary oedema or cardiogenic shock
* The investigator believes that the patient is not suitable to participate in the study or complete the follow-up prescribed by the protocol from other medical, social and psychological aspects
* The patient is currently participating in another randomized study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a prospective observational cohort study aimed at thoroughly investigating the disease progression and influencing factors of patients with moderate aortic valve disease, diagnosed at the Second Affiliated Hospital of Zhejiang University School of Medicine. Aortic valve stenosis and aortic regurgitation are the most common forms of aortic valve disease. According to the 2021 ESC guidelines, moderate aortic stenosis (Moderate AS) is defined as an aortic valve area (AVA) of 1.0-1.5 cm2 on echocardiography (or AVA &lt;1.0 cm2 with an AVA index of 0.60-0.85 cm2/m2), a peak jet velocity (Vmax) of 3-4 m/s, and/or a mean transvalvular gradient of 20-40 mmHg. Moderate aortic regurgitation (Moderate AR) is defined as a regurgitant fraction between 30% and 50% or an effective regurgitant orifice area between 0.10-0.30 cm2.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2034-01 (Estimated); Study Completion 2034-01 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 1-year, 3-year, and 5-year at follow-up
Re-hospitalization related to heart failure. | 1-year, 3-year, and 5-year at follow-up
Aortic valve replacement | 1-year, 3-year, and 5-year at follow-up
  Surgical Aortic Valve Replacement or Transcatheter Aortic Valve Replacement.
Stroke | 1-year, 3-year, and 5-year at follow-up
  Episode of ischemic stroke or hemorrhagic stroke in the internal carotid artery territory defined on CT scan or MRI brain.

SECONDARY OUTCOMES:
Change in echocardiography examination | 1-year, 3-year, and 5-year at follow-up
  valvular mean gradient
Change in cardiac CT examination | 1-year, 3-year, and 5-year at follow-up
  Calcium volume or calcium volume
Change in laboratory examination | 1-year, 3-year, and 5-year at follow-up
  elevation of pro-BNP levels

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Wang, Dorctor, Principal Investigator — Second Affiliated Hospital of Zhejiang University, School of Medicine
Locations (1):
- Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No